CLINICAL TRIAL: NCT00962273
Title: The Pandemic Stress Vaccine: Randomized Controlled Trial of an Educational Resource to Enhance the Resilience of Healthcare Workers Facing an Infectious Outbreak
Brief Title: The Pandemic Stress Vaccine: A Resource to Enhance the Resilience of Healthcare Workers Facing an Infectious Outbreak
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low participation and retention rates
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Dr. William Lancee - Head of Research, Department of Psychiatry, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09-0133-E
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Psychological Stress
Keywords: health personnel; communicable diseases; stress, psychological; resilience, psychological; disaster planning; education; online
MeSH Terms: conditions — Stress, Psychological; Communicable Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pandemic Stress Vaccine - Interactive (Experimental)
  Interventions: Behavioral: Interactive computerized learning resource
- Pandemic Stress Vaccine - Didactic (Active Comparator)
  Interventions: Behavioral: Didactic computerized learning resource
- Wait list (No Intervention): Some participants are assigned to an eight week waiting condition prior to the course commencing.

INTERVENTIONS:
Behavioral: Interactive computerized learning resource — In a series of interactive scenarios, participants can "see" themselves in stressful work situations that could arise during an influenza pandemic and reflect on effective ways to work out personal and interpersonal difficulties.
  Arms: Pandemic Stress Vaccine - Interactive
Behavioral: Didactic computerized learning resource — In a non-interactive format (i.e., a series of audio presentations with accompanying PowerPoint-type slides) participants are given information on how to handle stressful work situations that could arise during an influenza pandemic.
  Arms: Pandemic Stress Vaccine - Didactic

SUMMARY:
The purpose of this study is to determine the effects of an interactive, computerized learning resource designed to increase resilience in hospital-based health care workers preparing for an influenza pandemic. The effects of the learning resource will be compared to a non-interactive learning resource condition and a control condition. It is hypothesized that (a) online pandemic-related education reduces absenteeism and interpersonal problems for healthcare workers (HCWs), and improves their pandemic self-efficacy in the short and long-term, and (b) an interactive format for online education is necessary for its benefits.

ELIGIBILITY:
Inclusion Criteria:

* employee or professional staff of a hospital

Exclusion Criteria:

* unable to read and write English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Absenteeism | 32 weeks

SECONDARY OUTCOMES:
Pandemic self-efficacy | 32 weeks
Interpersonal problems | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William J. Lancee, Ph.D., Principal Investigator — MOUNT SINAI HOSPITAL; Robert G. Maunder, M.D., Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Maunder RG, Lancee WJ, Balderson KE, Bennett JP, Borgundvaag B, Evans S, Fernandes CM, Goldbloom DS, Gupta M, Hunter JJ, McGillis Hall L, Nagle LM, Pain C, Peczeniuk SS, Raymond G, Read N, Rourke SB, Steinberg RJ, Stewart TE, VanDeVelde-Coke S, Veldhorst GG, Wasylenki DA. Long-term psychological and occupational effects of providing hospital healthcare during SARS outbreak. Emerg Infect Dis. 2006 Dec;12(12):1924-32. doi: 10.3201/eid1212.060584. PMID 17326946